CLINICAL TRIAL: NCT05020613
Title: Comparison of Early and Late Removal of the Urinary Catheter After Low Anterior Resection
Brief Title: Early and Late Removal of the Urinary Catheter After Rectum Resection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Tevfik Kivilcim Uprak, MD, Marmara University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 412
Record Dates: First submitted 2021-08-19; First posted 2021-08-25 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Colorectal Surgery; Rectal Cancer; Urinary Retention Postoperative
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early group (Other): Patients whose catheters are removed within the first 48 hours after surgery will form the early group.
  Interventions: Procedure: Procedure: Early removal group
- Late group (Other): Patients whose catheters are removed after the first 48 hours of surgery will form the early group.
  Interventions: Procedure: Procedure: Late removal group

INTERVENTIONS:
Procedure: Procedure: Early removal group — Participants assigned this arm will have their urethral catheters removed at 2 days after low anterior resection of the rectum
  Arms: Early group
Procedure: Procedure: Late removal group — Participants assigned this arm will have their urethral catheters removed after 48.th hours after Low anterior resection of the rectum
  Arms: Late group

SUMMARY:
It was aimed to investigate the need for urinary retention and recatheterization in the postoperative period by removing the urinary catheter in patients undergoing low anterior resection, in the early or late period.

DETAILED DESCRIPTION:
Urinary catheter is placed before abdominal surgery to increase visualization during the operation, prevent bladder injury and provide perioperative urine output monitoring. It is especially useful in patients who will undergo low anterior resection, with a high risk of nerve damage and consequent urinary retention and bladder dysfunction. Urinary catheter removal time differs between operations. Traditionally, the urinary catheter is kept in place for 7 days because urinary retention occurs in some patients whose urinary catheter is displaced in the early period. As the urinary catheter retention time increases, the risk of urinary tract infection also increases.

According to the current ERAS protocol, it is recommended to remove the urinary catheter 48 hours after the surgery in patients who have undergone colorectal surgery and are treated with epidural pain management. However, the ERAS protocol is not specific to patients who have undergone low anterior resection, which is the main point of our study and includes all patients who have undergone colorectal surgery. Most authors still believe that prolonged retention of the urinary catheter will prevent urinary retention and long-term bladder dysfunction. In a randomized controlled study (published in 1999) that we encountered during our own literature search, early removal of the urinary catheter was associated with increased urinary retention [2]. In recent studies, some authors have associated the early removal of the urinary catheter with increased urinary retention [3], while others claimed the opposite and reported contradictory results [4]. Advances in laparoscopic techniques have made it possible to visualize the hypogastric and pelvic nerves (nerves associated with urinary functions) during surgery. In addition to these developments, dissections on embryonic planes and tumor reduction with neoadjuvant chemotherapy protect these nerves during surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients who will undergo Low Anterior Resection due to rectal cancer in the Department of General Surgery of our university.
* Competent to consent to participate in trial
* Elective surgery
* ASA classification of 1~3

Exclusion Criteria:

* Patients whose post-treatment status cannot be obtained.

  * Having Bladder surgery before
  * Having a previous prostate surgery.
  * Patient's refusal to participate in the study.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Post-operative urinary retention requiring re-catheterisation | 1 day
  Development of acute post-operative urinary retention requiring re-catheterisation within 1 day of removal of urethral catheter in the post-operative period.
Postoperative urine culture | 7 days
  Investigate any colonization before discharge in both groups
Discharge with urinary catheter | 7 days
  Any need for urinary catheter at the time of the discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara university Pendik Research and Education Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Duchalais E, Larson DW, Machairas N, Mathis KL, Dozois EJ, Kelley SR. Outcomes of Early Removal of Urinary Catheter Following Rectal Resection for Cancer. Ann Surg Oncol. 2019 Jan;26(1):79-85. doi: 10.1245/s10434-018-6822-x. Epub 2018 Oct 23. PMID 30353391
- [Background] Xu L, Tao ZY, Lu JY, Zhang GN, Qiu HZ, Wu B, Lin GL, Xu T, Xiao Y. A single-center, prospective, randomized clinical trial to investigate the optimal removal time of the urinary catheter after laparoscopic anterior resection of the rectum: study protocol for a randomized controlled trial. Trials. 2019 Feb 15;20(1):133. doi: 10.1186/s13063-019-3210-1. PMID 30770766
- [Background] Yoo BE, Kye BH, Kim HJ, Kim G, Kim JG, Cho HM. Early Removal of the Urinary Catheter After Total or Tumor-Specific Mesorectal Excision for Rectal Cancer Is Safe. Dis Colon Rectum. 2015 Jul;58(7):686-91. doi: 10.1097/DCR.0000000000000386. PMID 26200683